CLINICAL TRIAL: NCT03784105
Title: Effect of Codeine on Pharyngeal and Esophageal Motility in Healthy Subjects: a Double-blind, Placebo-controlled, Randomized, Cross-over Study
Brief Title: Codeine on Pharyngeal and Esophageal Motility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: S60496
Record Dates: First submitted 2018-12-11; First posted 2018-12-21 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Esophageal Motility Disorders
Keywords: codeine; Esophageal motility; Pharyngeal motility
MeSH Terms: conditions — Esophageal Motility Disorders | interventions — Codeine

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized, cross-over study in healthy volunteers
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind, preparation and administration of codeine or placebo conducted by an independent researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Codeine (Experimental)
  Interventions: Drug: Codeine Phosphate
- Siripus simplex (Placebo Comparator)
  Interventions: Drug: Siripus simplex

INTERVENTIONS:
Drug: Codeine Phosphate — 30 mL of codeine phosphate 10mg/5mL
  Arms: Codeine
Drug: Siripus simplex — Sugar syrup
  Arms: Siripus simplex

SUMMARY:
Opioids act on opioid receptors located in the brain as well as in the gastrointestinal (GI) tract to induce changes in motility. A variety of studies have linked chronic opioid use with changes in intestinal and to a lesser extent esophageal motility. Less is known about acute administration effects on distal esophageal motility and LES and even less with respect to proximal esophagus, UES and pharynx. Codeine, an opioid receptor agonist, by acting both centrally as well as in the periphery may induce changes in parts of the GI tract implicated in deglutition. Therefore, to evaluate the hypothesis the researchers will study motility patterns in the pharynx, UES, proximal and distal esophagus and LES in 22 healthy volunteers receiving placebo or codeine (60 mg) in a double-blind randomized cross-over controlled fashion. Motility patterns will be studied using state-of-the-art criteria and analytic tools (Chicago 3.0, AIMPlot analysis).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged between 18-60 years old
* Written informed consent

Exclusion Criteria:

* No chronic disease/medication
* No GI symptoms
* Not pregnant or breast-feeding
* No history of head/neck surgery
* Not allergic to codeine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Difference in distal contractile integral | 1 week
  The difference in distal contractile integral between the codeine and placebo condition
Difference in integrated relaxation pressure | 1 week
  The difference in integrated relaxation pressure between the codeine and placebo condition
Difference in distal latency | 1 week
  The difference in distal latency between the codeine and placebo condition.
Difference in pressure flow | 1 week
  The difference in pressure flow between the codeine and placebo condition

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Jan Tack, Leuven
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Geeraerts A, Geysen H, Ballet L, Hofmans C, Clevers E, Omari T, Manolakis AC, Mols R, Augustijns P, Vanuytsel T, Rommel N, Tack J, Pauwels A. Codeine induces increased resistance at the esophagogastric junction but has no effect on motility and bolus flow in the pharynx and upper esophageal sphincter in healthy volunteers: A randomized, double-blind, placebo-controlled, cross-over trial. Neurogastroenterol Motil. 2021 May;33(5):e14041. doi: 10.1111/nmo.14041. Epub 2020 Nov 24. PMID 33232555